CLINICAL TRIAL: NCT05330780
Title: Breathing Room Intervention to Achieve Better Lung Health in Older Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Milwaukee (Other)
Responsible Party: Principal Investigator, Murad Taani, Assistant Professor, University of Wisconsin, Milwaukee
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20.135
Record Dates: First submitted 2022-03-07; First posted 2022-04-15 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Breathing; Aging
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All participants (Experimental): The study will be single arm with intervention provided to all participants
  Interventions: Other: Breathing Room

INTERVENTIONS:
Other: Breathing Room — 8 total group classes performed twice a week over the course of 4 weeks, with IMTs utilized during the classes as well as 3 days outside of the class days at 5 sets of 5 breaths completed 5 times a day

SUMMARY:
This proposed study will evaluate whether a novel nonpharmacological intervention, Breathing Room, can improve lung function in the target population of older adults. Therefore, the primary aim of this pilot is to examine the effect of Breathing Room on inspiratory muscle strength, spirometry confirmed ventilatory function (Forced Expiratory Volume in one second (FEV1), Forced Vital Capacity (FVC) and FEV1/FVC), functional status, posture, physical activity, and lower respiratory infection rates.

DETAILED DESCRIPTION:
Restrictive ventilatory patterns (RVPs) contribute to two prevalent problems in older adults: 1) the development of pneumonia and other lower respiratory infections; and 2) declining endurance for physical activity. The Breathing Room was developed as an exercise activity designed to open the thoracic cage, increase strength of the muscles of respiration with inspiratory muscle trainers, and optimize the breathing technique.

This will be a pretest-posttest design in which the outcomes are measured at baseline, and at two weeks and four weeks post start of Breathing Room intervention. Breathing Room classes will be held 3 times a week for 4 weeks (2 group classes, 1 individual reinforcement of Inspiratory Muscle Training [IMT] homework). The IMT homework includes 3 days 5 cycles of 5 breaths, each cycle followed by 2-minute rest. The IMT will be also utilized during the 2 group classes.

The group classes will be conducted with a maximum of 5 participants in each group. Data on inspiratory muscle strength, spirometry confirmed ventilatory function (Forced Expiratory Volume in one second (FEV1), Forced Vital Capacity (FVC) and FEV1/FVC), functional status, posture, and physical activity will be collected. Infection rate data for each resident for 4 months following completion of Breathing Room will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* able to understand English
* baseline oxygen saturation level is above 85%
* spirometry-confirmed restrictive ventilatory pattern (forced vital capacity < 80% predicted, forced expiratory volume in 1 second/forced vital capacity ≥ 0.70

Exclusion Criteria:

* have lung disease classified as restrictive or obstructive
* have unstable angina/myocardial infarction, eye or lung surgery within the previous 8 weeks or aneurysm
* have had major orthopedic surgery in the last 12 weeks
* have been told they have heart failure, take a diuretic "water pill" and have been told to restrict their salt and fluid intake (symptoms that coincide with Stage C of heart failure based on the American College of Cardiology and the American Heart Association classification system
* score in the severely impaired range on the Short Orientation Memory Concentration Test
* history of spontaneous pneumothorax

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-02-22 (Actual); Primary Completion 2023-11-29 (Actual); Study Completion 2023-11-29 (Actual)

PRIMARY OUTCOMES:
Change in forced expiratory volume in one second (FEV1) | At baseline, after 2 weeks intervention, after 4 weeks intervention
  Spirometry testing will be performed using the MicroLoop battery operated portable spirometer to assess changes in forced expiratory volume in one second (FEV1) pre and post intervention
Change in inspiratory muscle strength | At baseline, after 2 weeks intervention, after 4 weeks intervention
  MicroRPM Respiratory Pressure Meter will be used to assess changes in inspiratory muscle strength pre and post intervention. The sniff nasal inspiratory pressure (SNIP) scores will be recorded pre and post intervention.
Change in functional capacity | At baseline, after 2 weeks intervention, after 4 weeks intervention
  The 6 Minute Walk Test will be used to assess the change in functional capacity and endurance pre and post intervention. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.
Change in grip Strength | At baseline, after 2 weeks intervention, after 4 weeks intervention
  A JAMAR hand dynamometer will be used to assess changes in grip strength pre and post intervention. Measurements will be recorded using participants' dominant and non-dominant hand and repeated 3 times to determine maximum grip strength.
Chane in kyphosis index | At baseline, after 2 weeks intervention, after 4 weeks intervention
  The flexicurve method will be used to measure the change in the kyphosis index pre and post intervention. To calculate the flexicurve kyphosis index, the apex kyphosis height (B) is divided by the length of the entire thoracic curve (X) and then multiplied by 100 (B/X × 100).
  The flexicurve ruler, which is a malleable band of metal covered with plastic and approximately 60 cm in length, will be used. The ruler can be bent in only one plane and retains the shape to which it is bent. The subject will be instructed to stand up straight and as tall as possible, and the flexicurve ruler will be aligned to the spine from C7 to T12. The ruler will be then placed flat on paper and its outline will be traced.
Change in forced vital capacity (FVC) | At baseline, after 2 weeks intervention, after 4 weeks intervention
  Spirometry testing will be performed using the MicroLoop battery operated portable spirometer to assess changes in forced vital capacity (FVC) pre and post intervention
Change in forced expiratory volume in one second/forced vital capacity (FEV1/FVC) ratio | At baseline, after 2 weeks intervention, after 4 weeks intervention
  Spirometry testing will be performed using the MicroLoop battery operated portable spirometer to assess changes in forced expiratory volume in one second/forced vital capacity (FEV1/FVC) ratio pre and post intervention

CONTACTS AND LOCATIONS:
Overall Officials: Murad H Taani, PhD, Principal Investigator — University of Wisconsin, Milwaukee
Locations (1):
- Ovation Communities (Jewish Home/Chai Point), Milwaukee, Wisconsin, United States